CLINICAL TRIAL: NCT07255352
Title: Investigation of the Effects of Suprahyoid Kinesio Taping on Swallowing Safety and Hyolaryngeal Elevation in Patients With Post-Stroke Dysphagia
Brief Title: Effect of Kinesio Taping Applied to the Suprahyoid Muscles on Swallowing Safety in Patients With Post-Stroke Dysphagia
Acronym: Post-Stroke KT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Omer Faruk Yasaroglu, Asst. Prof. Dr., Harran University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRÜ/24.14.41
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Dysphagia; Swallowing Disorder
Keywords: Kinesio Taping; Suprahyoid Muscles; Hyolaryngeal Elevation; Videofluoroscopic Swallowing Study
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Single group pre-test and post-test design. All participants receive Kinesio taping applied to the suprahyoid region, and swallowing parameters are evaluated before and after intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kinesio Taping Group (Experimental): Participants with post-stroke dysphagia will receive Kinesio Taping applied to the suprahyoid muscle region. Swallowing safety and kinematic parameters will be evaluated before and after the intervention.
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping — Kinesio tape will be applied over the suprahyoid region to facilitate muscle activation.

SUMMARY:
Dysphagia is defined as a disorder that occurs during the process of food transfer, beginning with oral intake and continuing until it reaches the stomach. The incidence of post-stroke dysphagia has been reported to range between 42% and 75%. Dysphagia can lead to aspiration pneumonia due to food entering the lungs, as well as malnutrition, dehydration, and even death. In patients with inadequate swallowing safety and efficiency, compensatory maneuvers such as chin tuck, head flexion, supraglottic swallowing, and the Mendelsohn maneuver are commonly used. These maneuvers aim to maintain oral intake by narrowing the laryngeal vestibule or increasing hyolaryngeal elevation. They are evaluated during videofluoroscopic swallowing studies and recommended to patients if they are found to prevent aspiration or penetration.

Kinesio taping (KT) has been reported to stimulate cutaneous receptors, increase sensory input, and facilitate neural reflexes, thereby promoting the activation of a greater number of motor units during maximal muscle contraction. In recent years, it has also begun to be used in the field of dysphagia rehabilitation. Studies conducted in stroke patients have shown that KT applied to the infrahyoid muscles provides resistance to the suprahyoid muscles and enhances their strength. A kinematic analysis study in stroke patients reported that KT applied to include the suprahyoid muscles increased vertical hyoid movement, although it did not result in a significant improvement in swallowing safety. The study, however, did not specify the detailed taping method used. Since the suprahyoid muscles are primarily responsible for hyolaryngeal elevation, KT focusing on this region has the potential to serve as a compensatory maneuver in dysphagia management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* Age over 18 years
* Presence of swallowing disorder symptoms
* Willingness to participate in the study

Exclusion Criteria:

* Presence of neurological diseases other than stroke
* Presence of tracheostomy
* Open wounds on the skin in the submental region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Swallowing Safety (Penetration-Aspiration Scale Score) | Immediately before and immediately after Kinesio taping application.
  Swallowing safety will be evaluated using the Penetration-Aspiration Scale (PAS) during videofluoroscopic swallowing study (VFSS). Each swallow will be scored on an 8-point scale, with higher scores indicating a higher risk of airway invasion. The difference in PAS scores before and immediately after Kinesio taping will be analyzed to assess the acute effect of the intervention on swallowing safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No